CLINICAL TRIAL: NCT04082520
Title: A Prospective, Phase II Study of Lutetium Lu 177 Dotatate (LUTATHERA®) in Patients With Inoperable, Progressive Meningioma After External Beam Radiation Therapy
Brief Title: Lutathera for the Treatment of Inoperable, Progressive Meningioma After External Beam Radiation Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1891; NCI-2019-05848 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1891 (Other: Mayo Clinic in Rochester); 17-009927 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Grade 1 Meningioma; Grade 2 Meningioma; Grade 3 Meningioma; Recurrent Meningioma; Unresectable Meningioma
MeSH Terms: conditions — Meningioma | interventions — Ga(III)-DOTATOC; gallium Ga 68 dotatate; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy; Specimen Handling; X-Rays; Photons

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (gallium Ga 68-DOTATATE PET/MRI, Lutathera) (Experimental): Patients receive gallium Ga 68-DOTATATE IV and undergo a PET/MRI or PET/CT before cycles 1 and 4. Patients then receive lutetium Lu 177 dotatate IV over 30-40 minutes. Treatment repeats every 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo MRI on study and during follow-up, as well as blood sample collection and possible SEPCT/CT dosimetry on study.
  Interventions: Radiation: Gallium Ga 68-DOTATATE; Drug: Lutetium Lu 177 Dotatate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Computed Tomography; Procedure: Biospecimen Collection; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Radiation: Gallium Ga 68-DOTATATE — Given IV
  Other Names: (68)Ga-DOTA-TATE; 68Ga-DOTA-0-Tyr3-Octreotate; 68Ga-DOTATATE; Gallium Ga 68 Oxodotreotide; Gallium Oxodotreotide Ga-68; Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Other: Questionnaire Administration — Ancillary studies
Procedure: Computed Tomography — Undergo PET/CT and/or SPECT/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography (CAT); computed axial tomography; computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT SCAN; tomography
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This phase II trial studies how well lutathera works in treating patients with meningioma that cannot be treated with surgery (inoperable) and is growing, spreading, or getting worse (progressive) after external beam radiation therapy. Lutathera is a radioactive drug administered in the vein that is designed to target and kill tumor cells. The goal of this study is to determine whether this drug is safe and effective in treating meningiomas that progress after radiation treatment. WHO Grade I and Cohort WHO II/III cohorts will be evaluated.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the efficacy of lutetium Lu 177 dotatate (LUTATHERA) treatment in patients with recurrent grade 1 meningioma as measured by 6-month progression-free survival (PFS) rate.

II. To estimate the efficacy of LUTATHERA treatment in patients with recurrent grade 2 or 3 meningioma as measured by 6-month PFS rate.

SECONDARY OBJECTIVES:

I. To determine the overall survival (by grade cohort) of patients with recurrent meningioma during or after treatment of LUTATHERA.

II. To determine the progression-free survival (by grade cohort) of patients with recurrent meningioma during or after treatment of LUTATHERA.

III. To determine the toxicity of LUTATHERA treatment in patients with recurrent meningioma.

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess the impact of treatment on the patient's quality of life (QOL) using the Promise-10, Brief Fatigue Inventory (BFI), and Mayo Patient Survey National Comprehensive Cancer Network (NCCN)-Functional Assessment of Cancer Therapy (FACT) Brain Symptom Index Questionnaire-24 (FBrSI-24) (version 2) instruments.

II. To compare the response assessment between standard of care brain magnetic resonance imaging (MRI) and gallium Ga 68-DOTATATE (68Ga-DOTATATE) positron emission tomography (PET) imaging.

III. To determine the best objective response (Macdonald criteria) of patients with recurrent meningioma during or after treatment of LUTATHERA.

IV. To determine the duration of local control with death as a competing risk (by grade cohort) of patients with recurrent meningioma during or after treatment of LUTATHERA.

V. To perform a quantitative dosimetric analysis of radiation dose delivered with lutathera:

Va. To determine intratherapeutic dosimetry for the target meningioma; Vb. To correlate treatment response of lutathera with target dose received; Vc. To determine intratherapeutic dosimetry for kidneys and other abdominal organs.

OUTLINE:

Patients receive gallium Ga 68-DOTATATE intravenously (IV) and undergo a PET/MRI or PET/computed tomography (CT) before cycles 1 and 4. Patients then receive lutetium Lu 177 dotatate IV over 30-40 minutes. Treatment repeats every 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo MRI on study and during follow-up, as well as blood sample collection and possible single photon emission computed tomography (SPECT)/CT dosimetry on study.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Previous treatment for meningioma including surgery, when possible, and radiation therapy (conventional fractionated or radiosurgery). Pathologic confirmation of meningioma is not required for patients who are not surgical candidates and received radiation therapy based on magnetic resonance imaging (MRI) consistent with meningioma. Patients with prior surgery will have pathologic confirmation of meningioma with either formalin-fixed paraffin-embedded (FFPE) tumor block OR meningioma tissue slides available for submission to central pathology review
* Radiographic evidence of meningioma progression with measurable disease, defined as an increase in size of the measurable primary lesion on imaging by 15% or more (sum of the bidirectional measurements) in an approximate 6 month time period (i.e., calculated rate of growth 15% / 6 months based on available scans) or by the appearance of a new measurable lesion
* Previous treatment with either fractionated radiation therapy or stereotactic radiosurgery at the site of progressive meningioma, without safe option for further radiotherapy
* Willing to undergo 68Ga-DOTATATE PET imaging. 68Ga-DOTATATE PET imaging must be Krenning score must be a score of 2 or higher, suggesting somatostatin receptor expression, to be registered on the study. A PET/MRI is preferred, but PET/CT is permitted if a patient is not technically able to receive a PET/MRI or at the discretion of the primary investigator (PI).
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2
* Absolute neutrophil count (ANC) >= 1500/mm (obtained =< 28 days prior to registration)
* Platelet count >= 100,000/mm (obtained =< 28 days prior to registration)
* Hemoglobin >= 9.0 g/dL (obtained =< 28 days prior to registration)
* Direct bilirubin < 1.5 x upper limit of normal (ULN) (or total bilirubin =< 3.0 x ULN with direct bilirubin =< 1.5 x ULN in patients with well-documented Gilbert's syndrome) (obtained =< 28 days prior to registration)
* Aspartate transaminase (AST) =< 3 x ULN (obtained =< 28 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulants (obtained =< 28 days prior to registration)
* Calculated creatinine clearance must be >= 40 ml/min using the Cockcroft-Gault formula (obtained =< 28 days prior to registration) using the Chronic Kidney Disease Epidemiology Collaboration (CDK-EPI) equation.
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study) and it is highly recommend to see study staff in Radiation Oncology, Medical Oncology and/or Neuro-Oncology during the Event Monitoring Phase of the study.
* Until 21 SPECT/CT slots are filled, willing to undergo SPECT/CT imaging for dosimetry analysis.

Exclusion Criteria:

* Eligibility for surgical or radiation treatment with curative intent
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women (NOTE: Patients with surgical sterilization or who have been post-menopausal for at least 2 years are excluded form pregnancy testing, but this must be documented.)
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Contraindications to or intolerance of MRI
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] II, III, IV), unstable angina pectoris, uncontrolled diabetes mellitus (fasting blood glucose > 2 ULN), cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm

  * Note: This includes treatment with somatostatin LAR within 4 weeks prior to enrollment, or any patient receiving treatment with short-acting octreotide that cannot be interrupted for greater than 24 hours before treatment
* Other active malignancy =< 2 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Current spontaneous urinary incontinence making impossible the safe administration of LUTATHERA
* Untreated, refractory and/or symptomatic toxicity related to previous radiation therapy including radiation necrosis, radiation optic neuropathy, or radiation retinopathy
* Optic nerve sheath meningioma, extracranial meningioma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2031-01-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival - 6 months | At 6 months after starting treatment
  Defined as the number of evaluable patients not having progressive disease or death within six months of the first day of treatment.

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  Defined as the time from the first day of treatment to death due to any cause.
Progression free survival - overall | Up to 5 years
  Defined as the time from the first day of treatment to the earliest date documentation of disease progression.
Incidence of adverse events | Up to 24 months
  Will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of adverse event will be recorded for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W. Merrell, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials